CLINICAL TRIAL: NCT02378311
Title: A Multicentre Observational Case-controlled Feasibility Study: In Children Who Ride Bikes or Scooters, is the Risk of Sustaining a Serious Injury Greater When Metal Handlebar Ends Are Exposed Than When They Are Covered by Intact Grips?
Brief Title: Handlebar Grip Related Injury Prevention (GRIP) Study: Are Exposed Metal Handlebar Ends a Risk Factor for Injury?
Acronym: GRIP
Status: Completed | Type: Observational
Sponsor: Andrew Neilson (Other)
Collaborators: University Hospitals Bristol and Weston NHS Foundation Trust (Other); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Andrew Neilson, Clinical Research Fellow, Paediatric Surgery, Birmingham Women's and Children's NHS Foundation Trust
Organization: Birmingham Women's and Children's NHS Foundation Trust (Other)
Other Study IDs: GRIPS-F-V4.15; 139699 (Registry Identifier: IRAS project ID); 15/LO/0311 (Other: REC reference)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Injuries; Trauma; Wounds and Injuries; Children; Child
Keywords: Bike; Bicycle; Scooter; Handlebar
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Those satisfying the inclusion & exclusion criteria whose injury involved impact with the handlebar end who have sustained an injury more severe than a skin or subcutaneous tissue contusion from an end-on handlebar impact
- Controls: Those satisfying the inclusion & exclusion criteria in whom the handlebars were not implicated in the mechanism of injury

SUMMARY:
Cycling injuries are the 3rd most common mechanism of injury in 7-13 year olds[1]. Bicycle injuries have remained one of the commonest causes of paediatric abdominal trauma for over 60 years[2,3]. 15% of child cyclist injuries involve impact with a handlebar; two-thirds of those are abdominal injuries[4]. Handlebar impact is now the commonest mechanism of major paediatric abdominal injury[3]. Serious handlebar injuries often occur after apparently minor falls; they are not unique to riders performing stunts[5].

One small study found that the metal handlebar ends were often exposed on bikes of children sustaining severe abdominal injuries[6]. Most European safety standards do not test grip durability[7-10]. Day-to-day use can damage rubber grips, exposing the underlying metal handlebar tube.

This feasibility study aims to test the research methods that will be used in a subsequent nationwide multicentre study. The main study will investigate the association between injuries and handlebar grip condition.

Children attending study hospitals with any bicycle or kick scooter injury will be invited to participate. Parents of injured children will be invited to complete questionnaires regarding circumstances surrounding the injury and condition of the handlebar ends on the bike or scooter involved. Clinical information regarding the injury will also be collected. The handlebar end condition will be compared between children sustaining a handlebar end injury [Cases] and riders whose injury did not involve the handlebar [Controls].

If exposed handlebar ends are more prevalent amongst riders with handlebar end injuries, injury prevention strategies can focus on methods to prevent damage occurring to grips through day-to-day use. If no such association is found, prevention strategies can be focused elsewhere, such as on design of effective protective clothing.

Data collection for this feasibility study will occur between March 2015 and September 2015.

The Chief Investigator, Mr. Andrew Neilson, funds the feasibility study.

DETAILED DESCRIPTION:
Injuries are the most common cause of death of children aged 1-14 years in the European Union[11]. In the United States cyclist injuries are the 3rd most common mechanism of injury in 7-13 year olds, after motor vehicle collisions (MVC) and falls[1]. Bicycle injuries have remained one of the most common causes of paediatric abdominal trauma for over 60 years[2,3]. The vast majority (95-98%) of child cyclists admitted due to abdominal trauma are over 5 years old[2,3]. As with most mechanisms of injury, boys are injured more frequently than girls. Around three quarters of injured child cyclists are boys[12].

In a recent UK study, handlebar end impact was the mechanism that most frequently resulted in major intra-abdominal trauma in children. Impact with a handlebar end was implicated in 29% of cases. This was ahead of falls (20%), pedestrians (8%) and MVC occupants (8%)[3]. A study conducted in Australia found 15% of child cyclist injuries involved impact with a handlebar, and 10% of all child cyclist injuries were abdominal handlebar injuries[4]. A study in Philadelphia found that 8% of all paediatric bicycle-related trauma admissions involved handlebars impacting the abdomen resulting in an injury with an Abbreviated Injury Scale (AIS) score of 2 or greater[13].

The majority of handlebar injury case series reported in the literature relate to children's abdominal injuries. The peak incidence occurs between 6 and 14 years of age[4]. However, adults can also sustain serious handlebar related injuries[14-16] and 36% of all handlebar injured patients sustain only extra-abdominal injuries[4]. It is not just pedal cyclists who are at risk of these injuries. Incidents also involve non-motorized kick scooters, moto-cross bikes, motorbikes and quad bikes[3,4].

Crash investigations have found that serious handlebar injuries often occur after apparently minor incidents; they are not unique to riders performing stunts or those riding BMX bikes[5,6]. There is a typical sequence of events common to many of these handlebar injuries[5]. The child loses control of the bike and begins to fall. The front wheel rotates through 90 degrees so that it is perpendicular to the child's body. The child continues to fall forwards, landing on the upturned handlebar end.

Children's bikes and scooters often have damaged rubber grips with exposed metal handlebar ends. This occurs through day-to-day use. Each time the child drops their bike or scooter on its side, the handlebar end contacts the ground. When it does so, the metal tube inside the rubber grip cuts into that rubber. With time, a circle is cut from the rubber end, exposing the metal pipe within.

Handlebar end injuries can occur both when the handlebar ends are exposed and when they are intact. Two studies from the 1990s have looked at the condition of the handlebar end implicated in such injuries[5,6].

Acton et al published a series of 21 patients who reported handlebar impact as the cause of their injuries. Re-interview found that metal handlebar ends were exposed on bikes of all 10 children who sustained a major abdominal injury, whilst exposed handlebar ends were present on only one bike of 8 respondents with minor abdominal injuries[6].

Winston et al included detailed analysis on 4 riders who sustained serious abdominal injuries due to landing on a handlebar end. They found that these serious injuries occurred in 3 riders despite the presence of protective rubber covering on the handlebar ends. The rider who impacted an exposed metal handlebar end, however, had a particularly serious injury. He was a 6-year-old boy who sustained a life threatening liver laceration[5].

Identifying if there is an association between the condition of handlebar grips and the likelihood of sustaining an injury is the ultimate aim of the main GRIP study. This feasibility study aims to test the intended methodology prior to rolling out a nationwide multicentre study. The feasibility study will allow power calculations to be performed for the nationwide study. The primary outcome of the nationwide study will address whether children falling onto exposed metal handlebar ends are at a greater risk of sustaining an injury than those who fall onto handlebars with intact rubber grips. A sub-study will explore whether there is any relationship between injury severity and grip condition.

Our clinical experience tells us that serious handlebar injuries do occur even when handlebar grips are intact. The investigators also know through anecdotes that some riders fall onto their handlebar ends and never attend hospital because no injury or only a minor injury is sustained. The cases presenting to tertiary paediatric units represent the 'tip of the iceberg'. A study to accurately identify the number of children who fall onto a handlebar but do not present to hospital is unlikely to be feasible. This is why the investigators have designed a case-controlled study.

If the nationwide multicentre GRIP study rejects the null hypothesis, then the investigators can focus on passive injury prevention strategies relating to handlebar ends. There are two aspects that could easily be addressed by safety standards. Grip durability and grip end minimum diameter. Improved durability should reduce the number of bikes or scooters in circulation with exposed metal handlebar ends. Larger diameter ends distribute any end-on impact over a larger surface area and hence reduce the pressure exerted on the point of contact.

Currently only one of the many applicable European safety standards includes a drop test of handlebar grip durability[9]. This standard for BMX bikes was introduced in 2012. However, the drop test has not been included in the more recently published standard for Bicycles for Young Children[10].

A minimum grip diameter requirement has been included in the standard for Bicycles for Young Children. It specifies that handlebars shall be fitted with handlebar grips, and that such grips shall be of resilient material and shall have an enlarged and covered end not less than 40mm in diameter[10]. That standard applies only to bikes suitable for children up to around 5 years of age. There is no such minimum handlebar end diameter requirement applied to bicycles ridden by children over 5 years of age, or to kick scooters. These standards simply require the handlebar to be fitted with handgrips or end plugs[7-9].

If, however, the nationwide multicentre GRIP study accepts the null hypothesis, the investigators can focus handlebar-related injury prevention on more complex mechanical solutions such as steering limiters or compressible handlebar ends, and on design of effective protective clothing. Some of the secondary outcomes the investigators propose addressing will be useful if it is found that exposed handlebar ends are not a risk factor for this injury mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-15 years inclusive
* Presenting to either of the study hospitals for assessment or treatment
* Sustained an injury or suspected to have sustained an injury (i.e. AIS >=0)
* Due to an incident involving any non-motorized bicycle, tricycle or kick scooter

Exclusion Criteria:

* Incidents where the injured child was involved in a motor vehicle collision
* Incidents where the injured child was injured by another rider (e.g. injured child run over by a cyclist)
* Incidents involving a bicycle fitted with 'bull bars'
* Patients for whom neither parent / guardian is fluent in English (if the history is clear from a parent, the patient will be eligible for inclusion)
* If an eligible patient is dead on arrival the family will not be invited to participate, and they will not subsequently be contacted
* If an eligible patient dies during their admission, they will be withdrawn from further involvement in the study and the family will not be contacted

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children attending either one of two tertiary paediatric hospital emergency departments and paediatric surgical units in the United Kingdom.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  To demonstrate the feasibility of a study researching whether or not exposed handlebar ends are a risk factor for injury in child bike and scooter riders.

SECONDARY OUTCOMES:
Research methodology | 6 months
  To test the research methodology proposed for a future nationwide multicentre study.
Power calculation data collection | 6 months
  To collect data required to do power calculations for a future nationwide multi centre study:
  The percentage of riders who did impact the handlebar end.
  The ratio of recruited Cases to Controls.
  The percentage who don't know whether they impacted the handlebar end.
  The percentage who don't know which handlebar end they hit.
  The proportion of intact, damaged and exposed handlebar ends in each group.
  The percentage whose handlebar ends are both in the same condition.

OTHER OUTCOMES:
Number of Cases & Controls | 6 months
  The total number of eligible Cases & Controls identified in each department.
Recruitment | 6 months
  The number identified by recruitment step 1a, 1b and 1c.
  Number recruited by reminder letters.
  Number of recruited participants who are eligible.
  Number completing questionnaire Part 2 without need for reminder.
  Number who respond to SMS, email, telephone or postal reminders for questionnaire Part 2.
  Proportion of responses to questionnaire Part 2 completed online versus using paper questionnaire.
  Proportion of incomplete versus complete questionnaire datasets.
  Number invited to participate in a telephone interview (Part 3).
  Number consenting to that interview; qualitative reasons for non-participation.
  Number completing that interview.
Study acceptability | 6 months
  Qualitative feedback from participants about the acceptability and design of the study.
  Qualitative feedback from recruiters about their willingness to recruit potential participants, the acceptability and design of the study.
Use of photographs | 6 months
  What proportion upload photos of their handlebar ends using the online form.
  What proportion of those using the paper questionnaire Part 2 email photos.
  Can an investigator grade handlebar condition using photos submitted by participants? If so, what is the inter-observer agreement between the parent's assessment and that of the investigator using the photograph.
Design & resources | 6 months
  Assess and record where possible the workload and resources required in each department.
  Record staff questions to aid compilation of an FAQ document for the national study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Neilson, MBChB, MRCS, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracy ET, Englum BR, Barbas AS, Foley C, Rice HE, Shapiro ML. Pediatric injury patterns by year of age. J Pediatr Surg. 2013 Jun;48(6):1384-8. doi: 10.1016/j.jpedsurg.2013.03.041. PMID 23845634
- [Background] Bergqvist D, Hedelin H, Lindblad B, Matzsch T. Abdominal injuries in children: an analysis of 348 cases. Injury. 1985 Jan;16(4):217-20. doi: 10.1016/s0020-1383(85)80001-2. PMID 3967900
- [Background] Getting to grips with handlebar injuries: a call for collaboration to inform legislative change. British Association of Paediatric Surgeons Annual Congress, Bournemouth 2013.
- [Background] Nataraja RM, Palmer CS, Arul GS, Bevan C, Crameri J. The full spectrum of handlebar injuries in children: a decade of experience. Injury. 2014 Apr;45(4):684-9. doi: 10.1016/j.injury.2013.07.022. Epub 2013 Dec 8. PMID 24321415
- [Background] Winston FK, Shaw KN, Kreshak AA, Schwarz DF, Gallagher PR, Cnaan A. Hidden spears: handlebars as injury hazards to children. Pediatrics. 1998 Sep;102(3 Pt 1):596-601. doi: 10.1542/peds.102.3.596. PMID 9738182
- [Background] Acton CH, Thomas S, Clark R, Pitt WR, Nixon JW, Leditschke JF. Bicycle incidents in children--abdominal trauma and handlebars. Med J Aust. 1994 Mar 21;160(6):344-6. PMID 8133818
- [Background] BSI. BS EN 14766:2005. Mountain bicycles: Safety requirements and test methods. British Standards Institution; 2006.
- [Background] BSI. BS EN 14619:2005. Roller sports equipment and kick scooters: Safety requirements and test methods. British Standards Institution; 2005.
- [Background] BSI. BS EN 16054:2012. BMX bicycles: Safety requirements and test methods. British Standards Institution; 2012.
- [Background] BSI. BS EN ISO 8098:2014. Cycles. Safety requirements for bicycles for young children. British Standards Institution; 2014.
- [Background] EuroSafe, Injury Database, European Commission, Swansea University, KFV. Injuries in the European Union, Issue 4. Summary of injury statistics for the years 2008-2010. European Association for Injury Prevention and Safety Promotion (EuroSafe); 2013.
- [Background] Acton CH, Thomas S, Nixon JW, Clark R, Pitt WR, Battistutta D. Children and bicycles: what is really happening? Studies of fatal and non-fatal bicycle injury. Inj Prev. 1995 Jun;1(2):86-91. doi: 10.1136/ip.1.2.86. PMID 9346002
- [Background] Winston FK, Weiss HB, Nance ML, Vivarelli-O'Neill C, Strotmeyer S, Lawrence BA, Miller TR. Estimates of the incidence and costs associated with handlebar-related injuries in children. Arch Pediatr Adolesc Med. 2002 Sep;156(9):922-8. doi: 10.1001/archpedi.156.9.922. PMID 12197801
- [Background] Nehoda H, Hochleitner BW. Subcapsular liver haematomas caused by bar ends in mountain-bike crashes. Lancet. 1998 Jan 31;351(9099):342. doi: 10.1016/s0140-6736(05)78334-3. No abstract available. PMID 9652623
- [Background] Bohmer JH, Proust AF. Adult bicycle handlebar injury. Am J Emerg Med. 2006 Sep;24(5):624-5. doi: 10.1016/j.ajem.2005.12.022. No abstract available. PMID 16938607
- [Background] Neofytou K, Michailidou M, Petrou A, Loizou S, Andreou C, Pedonomou M. Isolated jejunal perforation following bicycle handlebar injury in adults: a case report. Case Rep Emerg Med. 2013;2013:678678. doi: 10.1155/2013/678678. Epub 2013 Aug 5. PMID 23984116